CLINICAL TRIAL: NCT03345953
Title: Randomized Double Blind Parallel Groups Sequential, Placebo Controlled, Trial Assessing the Efficacy and Safety of BP1.4979 in Restless Legs Syndrome (RLS)
Brief Title: Clinical Trial Assessing the Efficacy and Safety of BP1.4979 in Restless Legs Syndrome
Acronym: P13-04
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study facing recruitment difficulties related to stringent eligibility criteria
Sponsor: Bioprojet (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P13-04 / BP 1.4979; 2013-004884-30 (EudraCT Number)
Record Dates: First submitted 2017-11-09; First posted 2017-11-17 (Actual); Last update posted 2020-07-30 (Actual); Status verified 2020-07

CONDITIONS: Restless Legs Syndrome
MeSH Terms: conditions — Restless Legs Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BP 1.4979 (Experimental): 15 mg tablet BID
  Interventions: Drug: BP 1.4979
- Placebo (Placebo Comparator): Matching placebo tablet
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BP 1.4979 — Double blind versus placebo
  Arms: BP 1.4979
Drug: Placebo — Double blind versus placebo
  Arms: Placebo

SUMMARY:
This is a Group Sequential Test multicenter, randomized, double blind, placebo controlled phase II proof of concept trial with parallel groups to evaluate the efficacy and the safety of BP1.4979 15mg BID compared to placebo in RLS patients during 2 weeks double blind treatment.

ELIGIBILITY:
Inclusion Criteria:

* Males or females > or = to 18 years
* 18 kg/m2 ≤ BMI ≤ 35 kg/m2
* Diagnosis of idiopathic RLS based on medical history and the presence of the 5 RLS diagnostic criteria and a normal clinical examination

  1. An urge to move the legs usually but not always accompanied by, or felt to be caused by, uncomfortable and unpleasant sensations in the legs.
  2. The urge to move the legs and any accompanying unpleasant sensations begin or worsen during periods of rest or inactivity such as lying down or sitting.
  3. The urge to move the legs and any accompanying unpleasant sensations are partially or totally relieved by movement, such as walking or stretching, at least as long as the activity continues.
  4. The urge to move the legs and any accompanying unpleasant sensations during rest or inactivity only occur or are worse in the evening or night than during the day.
  5. The occurrence of the above features is not solely accounted for as symptoms primary to another medical or a behavioral condition.
* The condition is not better explained by another current sleep disorder, medical or neurological disorder, mental disorder, medication use, or substance use disorder.
* RLS severity score > or = to 21/40 and RLS occurring at least 3 times per week for 'de novo' patients or after RLS treatment wash-out.
* Periodic Limb Movements during Sleep index > 15 for 'de novo' patients or after RLS treatment wash out.
* Not taking or accepting to discontinue drug therapy or medication for RLS, antipsychotic medication, antidepressant including Selective Serotonin Reuptake Inhibitors (SSRIs) prescribed for at least 5 half-lives prior to randomization (e.g. fluoxetine, paroxetine, fluvoxamine, sertraline, citalopram, escitalopram, venlafaxine, milnacipran, duloxetine) and/or any other psychotropic medication benzodiazepine and/or anticonvulsivants (gabapentine, pregabaline) prescribed to relief RLS, for at least 5 half-lives prior to randomization and/or opiates.
* Females of child-bearing potential must use a medically accepted effective method of birth control, agree to continue this method for the duration of the study and be negative to serum pregnancy test performed at the screening visit. Females should not be breast-feeding. Males accept to use child conception prevention method for the whole duration of the study
* In the opinion of the investigator, the subject must have adequate support to comply with the entire study requirements as described in the protocol (e.g. transportation to and from trial site, self-rating scales, drug compliance, scheduled visits, etc).
* Patient must have voluntarily expressed willingness to participate in this study, understand protocol procedures and have signed and dated an informed consent prior to beginning any protocol required procedures.

Exclusion Criteria:

* Any significant psychiatric illness (schizophrenia, bipolar disorder, severe depression, dementia, obsessive compulsive disorder...) or mood disorder, assessed by the Beck Depression Inventory (BDI) (exclusion if > or = to 16 and/ or item G ≠ 0).
* Abnormal neurological examination, history or presence of chronic pain other than that associated with RLS. History of epilepsy or serious head injury. History of peripheral neuropathy.
* Clinically significant sleep apnea (Apnea Hypopnea Index >15), narcolepsy, parasomnia as an adult, circadian rhythm disorder, or secondary causes of RLS (e.g chronic renal failure/hemodialysis).
* Other active clinically significant illness, including unstable cardiovascular, or neoplasic pathology which could interfere with the study conduct or counter-indicate the study treatments, place the subject at risk during the trial or interfere with study assessments or compromise the study participation.
* Subject with a known history of long QTc syndrome (e.g. syncope or arrhythmia) or presenting any significant serious abnormality of the ECG (e.g. recent myocardial infarction), or QTcB interval strictly higher than 450 ms.
* Subject with moderate hepatic impairment (transaminases > 1.5 ULN) or with renal impairment (creatinine clearance < 90 mL/min) , or with any other significant abnormality in the physical examination or clinical laboratory results (e.g positive laboratory test for Hepatitis B surface antigen (HBsAg), or anti-HIV 1/2 or anti- HCV antibodies).
* Iron deficiency (ferritin < 50 µg/l).
* Known hypersensitivity to the tested treatment including active substance and excipients.
* Use of drugs likely to influence sleep architecture or motor manifestations during sleep prior to randomization without an appropriate wash-out period. These include neuroleptics, L-dopa, dopamine agonists, hypnotics, sedatives, anxiolytics, antidepressants, anticonvulsants, psychostimulant medications, steroids in the evening, barbiturates, benzodiazepine treatment and opiates to relief RLS.
* Patient taking any prescription drug containing amphetamines.
* Recent history (≤ 1 year) of alcohol or drug abuse, or current evidence of substance dependence or abuse as defined by DSM-IV criteria (Gebauer L, LaBrie R et al. 2010).
* Regular consumption of large amounts of xanthine-containing substances (i.e more than 5 cups of coffee or equivalent amounts of xanthine-containing substance per day).
* Patient participating in another study and the use of any investigational therapy within the 30 days prior to the entry in this study.
* Patient without any medical care insurance.
* Pregnant woman or a pregnancy detected with a positive serum pregnancy test performed at the screening visit or lactating female.
* Male patient who wants to conceive a child for the whole duration of the study.
* Patient under guardianship who cannot provide consent on his own.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2018-02-06 (Actual); Primary Completion 2020-04-29 (Actual); Study Completion 2020-04-29 (Actual)

PRIMARY OUTCOMES:
Periodic Limb Movements per hour of Sleep (PLMS index) | 2 weeks
  Measure of the difference from baseline (Randomization) to the end of the double blind treatment period in Periodic Limb Movements per hour of Sleep (PLMS index) measured with PolySomnoGraphy (PSG)

SECONDARY OUTCOMES:
IRLSRS (International Restless Legs Syndrome Rating Scale) | 2 weeks
  Difference in IRLSRS score measured at randomization and end double blind study.treatment period. IRLSRS is ranging from 0 (no symptoms) to 40 (very severe symptoms)
Periodic Limb Movement during Wakefulness (PLMW) | 2 weeks
  Difference in PLMW measured at randomization and end double blind study treatment period. The PLMW will be measured during a Suggested Immobilization Test (1-hour test) to evaluate the limb movements during wakefulness.
Safety assessed by AEs collection | Up to 3 weeks
  Safety and tolerability of BP 1.4979 as assessed by AEs collection

CONTACTS AND LOCATIONS:
Overall Officials: Imad Ghorayeb, MD, Principal Investigator — Hôpital Pellegrin
Locations (1):
- Clinical Neurophysiology Department - Hôpital Pellegrin, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No